CLINICAL TRIAL: NCT02365935
Title: Phase II Randomized Controlled Trial on the Safety and Efficacy of 4 Versus 6 Courses of Adjuvant Chemotherapy in Locally Advanced Cervical Cancer Patients Previously Treated With Neoadjuvant Chemotherapy Plus Radical Surgery
Brief Title: 4 Versus 6 Courses of Adjuvant Chemotherapy in LACC Patients Previously Treated With NACT Plus Radical Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Roberto Angioli, Roberto Angioli, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC/47 cbm
Record Dates: First submitted 2015-01-21; First posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Uterine Cervical Neoplasms
Keywords: adjuvant chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A to administer 4 cycles (Experimental): In Group A, all patients received 4 cycles of adjuvant chemotherapy every three weeks according to the scheme Cisplatin 100 mg/mq and Paclitaxel 175 mg/mq.
  Interventions: Procedure: Group A adjuvant chemotherapy; Drug: Cisplatin; Drug: Paclitaxel
- Group B to administre 6 cycles (Experimental): In Group B, all patients received instead 6 cycles of adjuvant chemotherapy every three weeks according to the same chemotherapic regimen.
  Interventions: Procedure: Group B adjuvant chemotherapy; Drug: Cisplatin; Drug: Paclitaxel

INTERVENTIONS:
Procedure: Group A adjuvant chemotherapy — In Group A, all patients received 4 cycles of adjuvant chemotherapy every three weeks according to the scheme Cisplatin 100 mg/mq and Paclitaxel 175 mg/mq.
  Other Names: 4 cycles
  Arms: Group A to administer 4 cycles
Procedure: Group B adjuvant chemotherapy — In Group B, all patients received 6 cycles of adjuvant chemotherapy every three weeks according to the scheme Cisplatin 100 mg/mq and Paclitaxel 175 mg/mq.
  Arms: Group B to administre 6 cycles
Drug: Cisplatin
Drug: Paclitaxel

SUMMARY:
The investigators primary outcome was to evaluate the effectiveness in term of Overall Survival (OS) and disease free interval (DFI) of two different platinum-based chemotherapic regimen (3 and 6 cycles) for treatment of Locally Advanced Cervical Cancer (LACC) (IB2-IIB) previously treated with Neoadjuvant Chemotherapy Plus Radical Surgery (NACT+RS).

The secondary outcome was to evaluate and compare safety, in term of toxicity profile, of the two treatment options.

DETAILED DESCRIPTION:
Between February 2007 to January 2013, all patients with diagnosis of LAAC referred to the Division of Gynecologic Oncology of the Campus Bio-Medico University of Rome, were eligible for this protocol. The institutional internal review board approved the study. Inclusion criteria were: I) Patients with squamous cell, adenosquamous or adenocarcinoma of the cervix; II) Stage IB2-IIB according to the International Federation of Gynecology and Obstetrics (FIGO); III) age between 18 and 75 years; IV) Eastern Cooperative Oncology Group (ECOG) performance status 0-2; V) normal cardiac and respiratory functions; VI) absence of secondary malignancies; VII) no previous surgical, chemotherapic and/or radiotherapic treatment for secondary malignancies VIII) informed consent obtained from the patient.Exclusion criteria included: I) histological confirmation of papillary serous, mucinous, clear cell, squamous cell, mixed and undifferentiated carcinoma of the uterus; II) abnormal hepatic function (transaminases > 2.5 x upper limit, serum bilirubin > 1,5 x upper limit); III) abnormal renal function (creatinine clearance <60 mL/min and/or serum creatinine>2.0 mg/100 mL) function; IV) abnormal bone marrow function (absolute neutrophil count <1,5 x 109/L or platelet count < 100 x 109/L or hemoglobin < 9 g/dL; V) severe or uncontrolled infection, other systemic diseases or mental illness; and VI) pregnant women. Clinical staging was performed according to the NCCN criteria, and included pelvic examination, cervical biopsy, abdomen-pelvis Computed Tomography, chest X-ray; examination under anesthesia, cystoscopy and/or proctoscopy if clinically indicated (National Comprehensive Cancer Network, Clinical Practicw Guidelines in Oncology. Cervical Cancer, Version 2.2015) All patients who met inclusion and exclusion criteria were enrolled and received 3 cycles of neoadjuvant chemotherapy (NACT) every three weeks according to the scheme Cisplatin 100 mg/mq and Paclitaxel 175 mg/mq.

Complete response was defined as complete disappearance of all clinically detect able disease, determined by 2 observations not less than 4 weeks apart. Partial response was recorded as ≥50% reduction in total tumor size, determined by 2 observations not less than 4 weeks apart. No response or stable disease was defined as <50% decrease in tumor size or <25% increase in the size of one or more measurable lesions. Progressive disease was defined >25% increase in size or the appearance of new lesions.

After NACT all patients with stable or progressive disease were excluded from the protocol, all others were underwent to bilateral systematic pelvic lymph node dissection, classical radical hysterectomy and bilateral salpingo-oophorectomy. Aortic lymphadenectomy, up to the level of the inferior mesenteric artery, was reserved to patients with pelvic node disease at intraoperative examination or finding of bulky aortic nodes at the time of surgery. In case of positive aortic nodes, hysterectomy was not performed, patients were excluded from the protocol and referred to radiation oncologists. Similarly patients who presented positive surgical margins or close vaginal margins (<0.5 mm) at final pathology, were excluded from the study and referred to radiotherapist. After surgery were randomly allocated to undergo 4 or 6 cycles of chemotherapy by using a predetermined computer-generated randomisation code. In Group A, all patients received 4 cycles of adjuvant chemotherapy every three weeks according to the scheme Cisplatin 100 mg/mq and Paclitaxel 175 mg/mq.In Group B, all patients received instead 6 cycles of adjuvant chemotherapy every three weeks according to the same chemotherapic regimen. Adjuvant chemotherapy started within 28 days after surgery. Follow-up procedures included physical examination and vaginal cytology every 3 months for 2 years, then every 6 months until the 5th year according the NCCN 2015 and total body CT.

Therefore in all patients in whom there was suspicion of relapse, the total body CT was anticipated.

To assess the sample size, in agreement with the investigators experience, the investigators estimated a 20% reduction of the toxicity profile for patients who received 4 cycles of adjuvant chemotherapy compared to those who received 6 cycles (11; 19). Considering a power of 80%, to detect a statistically significant difference (alpha = 0.5; P = 0.05 Long Rank Test), 100 patients were necessary for each treatment arm.

OS and DFS curves were estimated using the Kaplan-Meier method and differences were compared by use of the log-rank test.

The comparison of other variables between two groups was evaluated using the Mann-Whitney test, the chi-square test, Fisher test. Statistical significance was set at p <0.05.

DFS, OS and recurrence rate were analyzed only in those patients who completed the study protocol; toxicity profile of the two treatment groups, however, were statistically analyzed considering all patients randomized and enrolled in the study protocol after treatment with NACT + RS.

ELIGIBILITY:
Inclusion Criteria:

* patients with squamous cell, adenosquamous or adenocarcinoma of the cervix
* Stage IB2-IIB according to the Inyernational Federation of Gynecology and Obstetrics (FIGO)
* age between 18 and 75 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* normal cardiac and respiratory functions
* absence of secondary malignancies
* no previous surgical, chemotherapic and/or radiotherapic treatment for secondary malignancies
* informed consent obtained from the patient.

Exclusion Criteria:

* histological confirmation of papillary serous, mucinous, clear cell, squamous cell, mixed and undifferentiated carcinoma of the uterus
* abnormal hepatic function (transaminases > 2.5 x upper limit, serum bilirubin > 1,5 x upper limit)
* abnormal renal function (creatinine clearance <60 mL/min and/or serum creatinine>2.0 mg/100 mL) function
* abnormal bone marrow function (absolute neutrophil count <1,5 x 109/L or platelet count < 100 x 109/L or hemoglobin < 9 g/dL
* severe or uncontrolled infection, other systemic diseases or mental illness; and
* pregnant women. Clinical staging was performed according to the NCCN criteria, and included pelvic examination, cervical biopsy, abdomen-pelvis Computed Tomography, chest X-ray; examination under anesthesia, cystoscopy and/or proctoscopy if clinically indicated (National Comprehensive Cancer Network, Clinical Practicw Guidelines in Oncology. Cervical Cancer, Version 2.2015)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2007-02; Primary Completion 2013-01 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
overall survival | up to 6 years
  To evaluate the effectiveness in term of overall survival of two different platinum-based chemotherapic regimen (4 and 6 cycles) for treatment of LACC (IB2-IIB) previously treated with NACT+RS.

SECONDARY OUTCOMES:
safety:to evaluate and compare safety, in term of toxicity profile, of the two adjuvant treatment options. | up to 6 years
disease free interval | up to 6 years
  To evaluate the effectiveness in term of disease free interval of two different platinum-based chemotherapic regimen (4 and 6 cycles) for treatment of LACC (IB2-IIB) previously treated with NACT+RS.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Angioli, Professor, Principal Investigator — Campus Bio Medico of Rome
Locations (1):
- campus bio-medico of Rome, Rome, Italy